CLINICAL TRIAL: NCT04906265
Title: Assessing the Outcome of Rehabilitation After Hip Fracture With a Wearable Device
Brief Title: Rehab After Hip Fracture With Wearable Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Collaborators: Malmo Municipality, Sweden (Unknown)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00789
Record Dates: First submitted 2021-05-07; First posted 2021-05-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Fracture of Hip
Keywords: Fracture of hip; Postural sway; Balance; Rehabilitation; Wearable device
MeSH Terms: conditions — Hip Fractures | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention comprises of standard rehabilitation and continuous measures of body positions and movements 24 hour a day with an IMU. Standard rehabilitation comprises of home-visits by a PT, where an individualized rehabilitation plan is outlined together with the patient. The plan includes individually tailored functional exercises. The plan also includes individually tailored walking exercises, indoor and outdoor when possible. At each home visit, the PT provides feedback to the participant based on the data from the IMU, i.e. body positions (time spent in sitting, standing, lying down) and body movements (steps per day, step length, walking speed).
  Interventions: Other: Intervention
- Control (Active Comparator): Standard rehabilitation alone
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — The intervention comprises of standard rehabilitation and continuous measures of body positions and movements 24 hour a day with an IMU. Standard rehabilitation comprises of home-visits by a PT, where an individualized rehabilitation plan is outlined together with the patient. The plan includes individually tailored functional exercises. The plan also includes individually tailored walking exercises, indoor and outdoor when possible. At each home visit, the PT provides feedback to the participant based on the data from the IMU, i.e. body positions (time spent in sitting, standing, lying down) and body movements (steps per day, step length, walking speed, sideway deviation during walking)
  Arms: Intervention
Other: Control — Standard rehabiliation
  Arms: Control

SUMMARY:
A randomized control trial, including two intervention arms with different methods for rehabilitation after hip fracture, conducted among persons with the need of rehabilitation in their own home.

DETAILED DESCRIPTION:
The increase of the aging population challenges health care providers. Fragility, oste-oporosis, and impaired balance are some major risk factors for hip fracture, an injury causing morbidity, mortality, and loss of independent life. This study aims to study if adding continuous measures of body positions and movements 24 hours a day with an Inertial Measurement Unit (IMU) can, compared to standard rehabilitation alone, optimize rehabilitation after hip fracture. The study is designed as a randomized controlled trial. Patients with hip fracture that require rehabilitation at home, will be invited to participate in the study. Those who accept to participate will randomly be assigned to intervention- or control group. The intervention comprises standard rehabilitation and continuous measures of body positions and movements 24 hours a day with an IMU. Standard rehabilitation comprises of home-visits by a PT, where an individualized rehabilitation plan is outlined together with the patient. The plan includes individually tailored functional exercises. The plan also includes individually tailored walking exercises, indoor and outdoor when possible. At each home visit, the PT provides feedback to the participant based on the data from the IMU, i.e. body positions (time spent in sitting, standing, lying down) and body movements (steps per day, step length, walking speed, sideway deviation during walking). The control group receives standard rehabilitation only. The primary outcome is balance, in terms of postural sway measured with the IMU, and functional balance measured with the Functional Balance test for Geriatric patients, secondary outcomes are health-related quality of life, measured with the EQ5D, functional independence in everyday activities, measured with the Barthel Index, fear of falling, measured with the Falls Efficacy Scale International, satisfaction with rehabilitation, measured with a single question, and compliance to the intervention .

ELIGIBILITY:
Inclusion Criteria:

* patients with a hip fracture, living in Malmö, and who are unable to visit a rehabilitation facility and therefore request treatment at home. Another inclusion criterion is the ability to read and understand the Swedish language or the ability to understand information through an interpreter.

Exclusion Criteria:

* the presence of major neurological diseases that have an impact on balance and walk-ing ability; a diagnosed cognitive disease, or moderate to severe cognitive impairment as assessed by a physiotherapist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in postural sway | Baseline, through study completion, on average 3 months
  Medio-lateral and anterior-posterior sway measured with the IMU in mm/sec

SECONDARY OUTCOMES:
Change in functional independence i everyday activities | Baseline and after study completion, on average 3 months
  The Barthel Index, likert scale, 6 items graded 0, 5, 10, 2 items graded 0, 5 and 2 items graded 0, 5, 10, 15. 100 highest possible score (best)
Change in function | Baseline and after study completion, on average 3 months
  EQ5D5L index from 0 (dead) to 1 (best imaginable health)
Change in health-related quality of life | Baseline and after study completion, on average 3 months
  EQ5D visual analogue scale, graded from 0 (worst health) to 100 (best health)
Change in functional balance | Baseline and after study completion, on average 3 months
  the Functional Balance test for Geriatric patients, including 4 tasks graded between 0-6,
Change in fear of falling | Baseline and after study completion, on average 3 months
  the Falls Efficacy Scale International , (22), comprising 16 questions with four possible answers
Satisfaction with rehabilitation | After study completion, on average 3 months
  Measured with a single question if the person thinks their need of rehabilitation is provided for, with four possible answers
Compliance to the intervention | Through study completion, on average 3 months
  Measured with a single question on how much the participant has trained since the last home visit, with three possible answers

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, Principal Investigator — Lund University, Medical Faculty, Dep of Health Sciences
Locations (1):
- Community Rehabilitation, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
Charing individual data is not aloud according to Swedish law